CLINICAL TRIAL: NCT07036419
Title: A Clinical Study on Efficacy and Safety of Remimazolam for Intraoperative Sedation in Pediatric and Adolescent Patients
Brief Title: A Trial of Remimazolam for Intraoperative Sedation in Pediatric and Adolescent Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR7056-207
Record Dates: First submitted 2025-06-16; First posted 2025-06-25 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Operative Sedation of Pediatric; Operative Sedation of Adolescent Patients
MeSH Terms: interventions — Injections; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam Group (Experimental)
  Interventions: Drug: Remimazolam Tosilate for injection
- Propofol Group (Active Comparator)
  Interventions: Drug: Propofol Injection

INTERVENTIONS:
Drug: Remimazolam Tosilate for injection — Remimazolam Tosilate for injection.
  Arms: Remimazolam Group
Drug: Propofol Injection — Propofol injection.
  Arms: Propofol Group

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of Remimazolam for intraoperative sedation in pediatric and adolescent patients.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent.
2. Subjects requiring elective general anesthesia surgery.
3. Male or female.
4. Meet the weight standard.

Exclusion Criteria:

1. Pediatric patients scheduled for elective cardiothoracic, neurosurgical, or hepatic surgery.
2. Patients who are planned to receive any anesthetic techniques other than total intravenous anesthesia (TIVA) from entry into the operating room until the end of surgery, such as inhalational anesthesia, epidural anesthesia, or spinal anesthesia.
3. Patients with a medical history or clinical evidence that may increase the risk of sedation or anesthesia and are deemed unsuitable for participation by the investigator.
4. Patients with a history of asthma or with risk for difficult mask ventilation or difficult intubation by the investigator's judgment.
5. With clinically significant abnormal clinical laboratory test value.
6. Known intolerance or allergy to benzodiazepines, propofol, opioids, neuromuscular blocking agents, or any of their components.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 138 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
The overall sedation success rate. | Throughout the anesthesia procedure.
  The overall sedation success rate, which encompasses both successful induction of sedation and successful maintenance of adequate sedation throughout the anesthesia procedure.

SECONDARY OUTCOMES:
Proportion of subjects with hemodynamic instability. | Up to 2 days.
  Defined as a ≥ ±20% change from the baseline in blood pressure or heart rate.
Incidence and severity of adverse events during the study. | Up to 3 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Children's Medical Center Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided